CLINICAL TRIAL: NCT06492330
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Proof of Concept Study Evaluating the Efficacy, Safety, and Tolerability of CS0159 Combined With Semaglutide in MASH Patients With Obesity and T2DM
Brief Title: Efficacy and Safety of CS0159 Combined With Semaglutide in MASH Patients With Obesity and T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, PHD, MD, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MASH-CS0159-IIT
Record Dates: First submitted 2024-06-25; First posted 2024-07-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Dysfunction-Associated Steatohepatitis (MASH); Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4mg CS0159 (Active Comparator): 4mg CS0159 (oral, once daily) + 0.5mg Semaglutide (subcutaneous injection, once weekly) for 16 weeks
  Interventions: Drug: CS0159
- CS0159 Placebo (Placebo Comparator): CS0159 placebo (oral, once daily) + 0.5mg Semaglutide (subcutaneous injection, once weekly) for 16 weeks
  Interventions: Drug: CS0159 placebo

INTERVENTIONS:
Drug: CS0159 — The intervention will include a 2-week screening period, a 16-week treatment period, and a 4-week follow-up period. Efficacy and safety evaluations will be conducted after the end of the treatment. During the 16-week treatment period, subjects will receive 4mg CS0159 (oral, once daily) + 0.5mg Semaglutide (subcutaneous injection, once weekly).
  Arms: 4mg CS0159
Drug: CS0159 placebo — The intervention will include a 2-week screening period, a 16-week treatment period, and a 4-week follow-up period. Efficacy and safety evaluations will be conducted after the end of the treatment. During the 16-week treatment period, subjects will receive CS0159 placebo (oral, once daily) + 0.5mg Semaglutide (subcutaneous injection, once weekly).
  Arms: CS0159 Placebo

SUMMARY:
This is an exploratory study evaluating CS0159 in combination with Semaglutide in MASH patients with obesity and T2DM.

DETAILED DESCRIPTION:
This is an exploratory study to evaluate the efficacy, safety, and tolerability of CS0159 in combination with Semaglutide in MASH patients with obesity and T2DM. A total of 60 patients will be recruited. BMI ≥35 kg/m2 will be used as a randomized stratification factor, and patients will be randomly assigned in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age≥18 and ≤65 years, male or female.
* 2. Patients with previous liver biopsy for MASH or MRI-PDFF ≥10% within 3 months prior to randomization.
* 3. Diagnosis of T2DM.
* 4. HbA1c: 7.0%-10.5%.
* 5. FPG: 7.0-13.3 mmol/L.
* 6. BMI: 30-45 kg/m2.
* 7. Subjects control blood glucose only by lifestyle intervention for at least 3 months before the screening period.
* 8. Willing to maintain consistent diet and exercise habits throughout the entire study, and adhere to the study protocol for timely administration of the study drug, and timely self-monitoring of blood glucose and recording.

Exclusion Criteria:

* 1. ALT≥2.5×ULN, AST≥2.5×ULN, TBil≥2×ULN, creatinine (Cr) ≥1.5×ULN and Serum creatinine clearance<60 mL/min, PLT<100×10^9/L, INR >1.3, ALB <3.5 g/dL.
* 2. Use of glucose-lowering medication in the 3 months prior to randomization.
* 3. Weight loss ≥ 5% in the 3 months prior to randomization or ≥10% in the 6 months prior to randomization or use of other weight-lowering drugs, corticosteroids, and etc.
* 4. History of allergy to glucagon-like peptide-1 receptor agonists (GLP-1RA) medications, currently in an allergic state, having allergic conditions, or history of allergies to ≥2 substances.
* 5. Subjects with T1DM, monogenic diabetes, diabetes caused by pancreatic damage, or other secondary diabetes.
* 6. Subjects with a history of severe pruritus.
* 7. Uncontrolled and potentially unstable diabetic retinopathy or maculopathy.
* 8. Thyroid C-cell tumour or family history, multiple endocrine neoplasia type 2 or family history.
* 9. History of acute or chronic pancreatitis.
* 10. Subjects with Child-Pugh class B or C grade cirrhosis.
* 11. HBsAg positive, HCV Ab positive, HIV Ab positive, TP Ab positive.
* 12. Arrhythmias, male QTc≥450 ms, or female QTc≥470 ms. Or cardiovascular disease for which the researcher has assessed that participation in the trial is not appropriate.
* 13. Diseases that interfere with the absorption, distribution, metabolism or excretion.
* 14. Gastrointestinal diseases that affect food digestion and absorption.
* 15. Use moderate or strong inhibitors or inducers of cytochrome P450 enzyme (CYP3A4 enzyme) within the first 14 days of randomization and throughout the entire trial period.
* 16. History of malignant tumors within the first 5 years of randomization.
* 17. Serious hypoglycemic events occurring ≥ 3 times within 12 weeks prior to administration, or acute and severe metabolic disorder occurred within 12 weeks prior to administration.
* 18. Drug abuse or alcohol abuse within the first 6 months of randomization.
* 19. Poor blood pressure control.
* 20. Mental illness, epilepsy.
* 21. Patients with uncontrollable severe infectious diseases before randomization.
* 22. Pregnant, planned pregnancy or breastfeeding.
* 23. Participated in other clinical trials in the first three months of randomization.
* 24. Any condition that in the judgement of the researcher precludes participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight relative to baseline | Baseline to 16 weeks
  Evaluate the percentage change in body weight relative to baseline after 16 weeks of treatment.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Baseline to 16 weeks
  Safety outcomes
Patient Health Questionnaire 9 (PHQ-9) | Baseline to 16 weeks
  Safety outcomes
Short form 36 health survey questionnaire (SF-36) | Baseline to 16 weeks
  Safety outcomes
Visual analog scale for pruritus and 5-D itch scale | Baseline to 16 weeks
  Safety outcomes
Proportion of subjects achieving ≥5% weight loss | Baseline to 16 weeks
  Proportion of subjects achieving ≥5% weight loss from baseline after 16 weeks of treatment.
Percentage change in HbA1c relative to baseline | Baseline to 16 weeks
  Evaluate the percentage change in glycated hemoglobin (HbA1c) relative to baseline after 16 weeks of treatment.
Fasting plasma glucose levels | Baseline to 16 weeks
  Changes in fasting plasma glucose levels relative to baseline after 16 weeks of treatment.
2-hour post-prandial plasma glucose levels | Baseline to 16 weeks
  Changes in 2-hour post-prandial plasma glucose levels relative to baseline after 16 weeks of treatment.
Fasting serum insulin levels | Baseline to 16 weeks
  Changes in fasting serum insulin levels relative to baseline after 16 weeks of treatment.
2-hour post-prandial serum insulin levels | Baseline to 16 weeks
  Changes in 2-hour post-prandial serum insulin levels relative to baseline after 16 weeks of treatment.
Fasting serum C peptide levels | Baseline to 16 weeks
  Changes in fasting serum C peptide levels relative to baseline after 16 weeks of treatment.
2-hour post-prandial serum C peptide levels | Baseline to 16 weeks
  Changes in 2-hour post-prandial serum C peptide levels relative to baseline after 16 weeks of treatment.
Percentage change in liver fat content relative to baseline | Baseline to 16 weeks
  Evaluate the percentage change in liver fat content measured by Magnetic resonance imaging-proton density fat fraction (MRI-PDFF) relative to baseline after 16 weeks of treatment.
Changes relative to baseline in body mass index (BMI) | Baseline to 16 weeks
  Changes in BMI (=body weight/height^2) relative to baseline after 16 weeks of treatment.
Changes relative to baseline in body composition | Baseline to 16 weeks
  Changes in body composition relative to baseline after 16 weeks of treatment, including lean mass, fat mass, body fat percentage and etc.
Changes relative to baseline in waist circumference and waist-to-hip ratio (WHR) | Baseline to 16 weeks
  Changes in waist circumference and waist-to-hip ratio (=waist circumference/hip circumference) relative to baseline after 16 weeks of treatment.
Changes relative to baseline in liver function | Baseline to 16 weeks
  including alanine aminotransferase, aspartate aminotransferase，ɣ-glutamyltransferase, alkaline phosphatase, lactate dehydrogenase, total bilirubin, direct bilirubin, total protein, albumin, and total bile acid.
Changes relative to baseline in renal function | Baseline to 16 weeks
  including including serum urea nitrogen, serum creatinine, and serum urinary acid.
Changes relative to baseline in lipid profile | Baseline to 16 weeks
  including serum triglycerides, total cholesterol, low-density lipoprotein cholesterol and high-density lipoprotein cholesterol.
Changes relative to baseline in parameters of hepatic fibrosis | Baseline to 16 weeks
  including serum hyaluronic acid, laminin, procollagen type III, and collagen type IV.

CONTACTS AND LOCATIONS:
Locations (1):
- Dep.endocrinology of Shanghai Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China